CLINICAL TRIAL: NCT01446445
Title: Individualization of Ganciclovir and Valganciclovir Doses in Renal Transplant Patients for Prophylaxis or Treatment of Cytomegalovirus(CMV)Infection Using Bayesian Prediction.
Brief Title: Individualization of Ganciclovir and Valganciclovir Doses Using Bayesian Prediction in Renal Transplant Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nuria Lloberas (Other)
Collaborators: Ministerio de Sanidad, Servicios Sociales e Igualdad (Other Government)
Responsible Party: Sponsor-Investigator, Nuria Lloberas, Clinical Investigator of Nephrology Department, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCV2010; 2010-021433-32 (EudraCT Number)
Record Dates: First submitted 2011-09-19; First posted 2011-10-05 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Infection in Solid Organ Transplant Recipients
Keywords: Cytomegalovirus; renal transplant
MeSH Terms: interventions — Ganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1.A (Prophylaxis-SPC) (Active Comparator): Prophylaxis for CMV infection and Ganciclovir/ Valganciclovir doses according to summaries of product characteristics (SPC).
  Interventions: Drug: Ganciclovir/ Valganciclovir according to SPC
- 1.B (Prophylaxis- PK model) (Experimental): Prophylaxis for CMV infection and Ganciclovir/Valganciclovir doses according to pharmacokinetic model.
  Interventions: Drug: Ganciclovir/ Valganciclovir according to PK model
- 2.A (Treatment-SPC) (Active Comparator): Treatment for CMV infection/disease and Ganciclovir/ Valganciclovir doses according to summaries of product characteristics (SPC).
  Interventions: Drug: Ganciclovir/ Valganciclovir according to SPC
- 2.B (Treatment-PK model) (Experimental): Treatment for CMV infection/disease and Ganciclovir/Valganciclovir doses according to pharmacokinetic model
  Interventions: Drug: Ganciclovir/ Valganciclovir according to PK model

INTERVENTIONS:
Drug: Ganciclovir/ Valganciclovir according to SPC — Doses according to Summaries of Product Characteristics (SPC)
  Other Names: Cymevene and Valcyte doses calculated according to SPC
  Arms: 1.A (Prophylaxis-SPC); 2.A (Treatment-SPC)
Drug: Ganciclovir/ Valganciclovir according to PK model — Doses according to population pharmacokinetic model
  Other Names: Cymevene and Valcyte doses calculated according to PK model
  Arms: 1.B (Prophylaxis- PK model); 2.B (Treatment-PK model)

SUMMARY:
The objective of the present study is to optimize intravenous ganciclovir(GCV) and oral valganciclovir (VGCV)doses, advised by the drug exposure, indicated by the area under the concentration time curve (AUC), in renal transplant patients receiving oral VGCV or intravenous GCV for CMV prophylaxis or treatment. The initial doses will be calculated according to population pharmacokinetic model. Subsequent doses will be adjusted according to plasma GCV concentrations, using the Bayesian approach. This method of dose adjustments could lead to increase the percentage of patients achieving a therapeutic exposure.

DETAILED DESCRIPTION:
The area under the concentration time curve of serum concentrations of GCV is an indicator of systemic exposure to the drug and is related to the effectiveness and safety. According to the population model developed by our group, less than 16% of patients treated achieve the therapeutic goal of AUC (40 to 50 mcg • h / L) after drug dosing according to summary of product characteristics (SPC). Especially, patients with impaired renal function values (creatinine clearance (CrC)l <30 ml / min) or high (CrCl> 70 ml / min) would be overdosed and underdosed, respectively, with the risk of more adverse effects or therapeutic failure.

Therefore, the individualization of the dosage of GCV, can contribute greatly to achieve optimal exposure to the drug in transplant patients, especially in the cases of extreme values of renal function (CrCl decreased and high). As a consequence, minimize adverse effects, ensure greater efficiency in the target population and reduce associated costs.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 or older, weigh more than 34kg and may be of either sex and race.
* Subjects must be willing to give informed consent (IC) in writing and be able to do and follow the study. If a subject cannot give informed consent in writing , a legal representative could sign in his place.
* Women of childbearing potential should perform a pregnancy test at the time of entry and accept the use of a medically acceptable contraceptive method during the study.

Exclusion Criteria:

* Creatinine Clearance (CrCl )<10 mL / min.
* Subjects may not have a history of type I hypersensitivity or idiosyncratic reactions to drugs ganciclovir/valganciclovir
* Pregnancy women.
* Women breast feeding
* Subjects may not present at time of inclusion any clinically significant disease that could interfere with study evaluations.
* Previous participation in another clinical trial sponsored by pharmaceutical industry, in which the promoter and the protocol set which should be the treatment for CMV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Area under the concentration time curve (AUC)of ganciclovir in steady state | Change from baseline to the end of the treatment, with an expected average of treatment of 4 weeks in treatment and 90 days in prophylaxis patients.
  Values of AUC of ganciclovir achieved with each intervention, that is, ganciclovir and valganciclovir dose adjustment according to SPC(specific product characteristics) or PK (pharmacokinetic) model.
  In each intervention: after starting treatment, change in route of administration, change in renal clearance >10 mL/min and end of treatment blood sampling for pharmacokinetic analysis will be performed in order to calculate AUC.

SECONDARY OUTCOMES:
CMV viral load measured by quantitative polymerase chain reaction (PCR) | Change from baseline to day 30 of study entry
  CMV viral load will be correlated with the exposure to ganciclovir during treatment period, in both interventions.
CMV viral load measured by quantitative polymerase chain reaction (PCR) | Change from baseline to day 60 of study entry
  CMV viral load will be correlated with the exposure to ganciclovir during treatment period, in both interventions.
CMV viral load measured by quantitative polymerase chain reaction (PCR) | Change from baseline to day 90 of study entry
  CMV viral load will be correlated with the exposure to ganciclovir during treatment period, in both interventions.
T-cell immune response against CMV infection measured by Enzyme-linked immunosorbent spot (ELISPOT) | Change from day 40 of treatment to day 20 after end of treatment.
  In prophylaxis patients(arm 1.A and 1.B): ELISPOT assay will be performed to assess the immune response to CMV viral infection on day 40 of initial dose and on day 20 after end of prophylactic therapy.
T-cell immune response against CMV infection measured by Enzyme-linked immunosorbent spot (ELISPOT) | Change from baseline to day 20 of treatment
  In treatment patients(arm 2.A and 2.B): ELISPOT assay will be performed to assess the immune response to CMV viral infection at baseline, day 10 and 20 of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nuria Lloberas, Ph.D, Principal Investigator — Nephrology Department-Hospital Universitari Bellvitge
Locations (1):
- Nephrology Department- Hospital Universitari Bellvtge, L'Hospitalet de Llobregat, Barcelona, Spain

REFERENCES:
- [Derived] Vernooij RW, Michael M, Colombijn JM, Owers DS, Webster AC, Strippoli GF, Hodson EM. Pre-emptive treatment for cytomegalovirus viraemia to prevent cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2025 Jan 14;1(1):CD005133. doi: 10.1002/14651858.CD005133.pub4. PMID 39807668
- [Derived] Vernooij RW, Michael M, Ladhani M, Webster AC, Strippoli GF, Craig JC, Hodson EM. Antiviral medications for preventing cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2024 May 3;5(5):CD003774. doi: 10.1002/14651858.CD003774.pub5. PMID 38700045
- [Derived] Padulles A, Colom H, Bestard O, Melilli E, Sabe N, Rigo R, Niubo J, Torras J, Llado L, Manito N, Caldes A, Cruzado JM, Grinyo JM, Lloberas N. Contribution of Population Pharmacokinetics to Dose Optimization of Ganciclovir-Valganciclovir in Solid-Organ Transplant Patients. Antimicrob Agents Chemother. 2016 Mar 25;60(4):1992-2002. doi: 10.1128/AAC.02130-15. Print 2016 Apr. PMID 26824942